CLINICAL TRIAL: NCT05079373
Title: Study of Neurological Damage From Coronavirus Disease (COVID-19): Extraction of Quantitative Imaging Biomarkers for the Characterization of Pathological Profiles
Brief Title: Study of Neurological Damage From Coronavirus Disease (COVID-19)
Acronym: NeuroBiomarK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8184
Record Dates: First submitted 2021-10-13; First posted 2021-10-15 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-COV-2; Central nervous system; Headache; Loss of smell; Coma
MeSH Terms: conditions — COVID-19; Headache; Anosmia; Coma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to support the exploration of the NEURO-COVID-19 database and in particular to carry out the post-treatments necessary to derive quantitative information on the characterization of the lesion load, in particular with regard to of the vascular tree

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years old)
* COVID + patient presenting with neurological symptoms leading to an MRI.
* Patient taken care of in one of the care centers associated with this research
* Patient not having expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Exclusion criteria:

* Patient who expressed his opposition to participating in the study
* COVID patient not having neurological symptoms or not having received an MRI
* Patient under guardianship or guardianship
* Patient under legal protection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient having covid and presenting with neurological symptoms leading to an MRI.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-10-09 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of the neurological damage in patients with Covid-19 | Files analysed retrospectively from January 01, 2020 to October 31, 2021 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Imagerie 2 - Neuroradiologie et Radiologie Ostéo-articulaire - Hôpitaux Universitaires de Strasbourg, Strasbourg, France